CLINICAL TRIAL: NCT05837078
Title: Effect of Laser Bio-stimulation on Peri-implant Tissue Health for Mandibular Knife-edge Ridges Managed With One- Stage Ridge Splitting and Two- Implant Mandibular PEEK Overdentures. A One -Year Randomized Controlled Trial
Brief Title: Effect of Laser Biostimulation With Mandibular Ridge Splitting and Peek Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Marwa adel, assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01100918
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Ridge Splitting
Keywords: peek , laser

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): patients had ridge splitting without laser bio stimulation and received two implants supported peek overdenture
  Interventions: Procedure: ridge splitting with implant placement
- study group (Active Comparator): patients had ridge splitting with laser bio stimulation and received two implants supported peek overdenture
  Interventions: Procedure: ridge splitting with implant placement

INTERVENTIONS:
Procedure: ridge splitting with implant placement — ridge splitting of mandibular denture followed by two implant placement

SUMMARY:
This study was conducted to determine the effectiveness of two-implant retained polyetheretherketone (PEEK) overdentures on reducing the transmitted forces on implants placed with ridge splitting either treated with laser biostimulation or not.

DETAILED DESCRIPTION:
This randomised controlled trial was executed on 18 completely edentulous patients from the Outpatient Clinic of the Faculty of Dentistry at Mansoura University in Egypt.

ELIGIBILITY:
Inclusion Criteria:

- eligible patients must have mandibular knife edge ridge

Exclusion Criteria:

* contraindicated any systemic disease preventing surgical intervention such as bone metabollic disease , diabetes mellitus

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
crestal bone loss | one year
  measuring marginal bone loss arround dental implants in mm by digital radiograph
plaque index | One year
  score 0 = no plaque; score1 = plaque only detected with a probe; score 2 = plaque visible to the naked eye; score 3 = abundant plaque1111
bleeding index | one year
  score 0: no bleeding when using a periodontal probe; score1: isolated bleeding spots visible; score 2: a confluent red line of blood along the mucosal margin; score 3: heavy or profuse bleeding).
gingival index | one year
  Score 0: normal peri implant mucosa; score 1: mild inflammation, slight colour change, and slight edoema; score 2: moderate inflammation, redness, edoema, and glazing; and score 3: severe inflammation, marked redness and edoema, and ulceration.
probing depth | one year
  A periodontal probe was used to measure pocket depth (PD). The distance between the marginal border of the mucosa and the tip of the periodontal probe at the base of the gingival sulcus was scored as the probing depth.

CONTACTS AND LOCATIONS:
Overall Officials: marwa adel, MD, Principal Investigator — Mansoura University
Locations (1):
- Marwa Adel, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No